CLINICAL TRIAL: NCT05712733
Title: Cholecystitis From a Microbiological and Histopathological Perspective
Status: Recruiting | Type: Observational
Sponsor: Organkirurgisk afdeling, sygehus lillebælt, Kolding (Network)
Responsible Party: Principal Investigator, Malene Borgager Dissing, Malene Børgager Dissing, MD, Organkirurgisk afdeling, sygehus lillebælt, Kolding
Other Study IDs: MBDissing
Record Dates: First submitted 2023-01-16; First posted 2023-02-03 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: Calculous Cholecystitis; Antibiotic Resistant Infection; Gallbladder Inflammation
MeSH Terms: conditions — Cholecystitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 14 Days
Biospecimen Retention: Samples With DNA — For microbiological analysis: bile fluid and gallbladder wall specimens For histopathologiical investigation: the gallbladder
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case group: Patients suffering from acute calculous cholecystitis undergoing subacute laparoscopic cholecystectomy.
  Samples of bile and gallbladder wall specimens will be taken during surgery and will be sent for microbiological and pathological investigation
  Interventions: Other: Microbiological and histopathological investigation of bile and gallbladder wall specimens.
- Control group: Patients suffering from painattacks due to gallstones, who have not symptoms of cholecystitis. The patients will undergo elective laparoscopic cholecystectomy.
  Samples of bile and gallbladder wall specimens will be taken during surgery and will be sent for microbiological and pathological investigation
  Interventions: Other: Microbiological and histopathological investigation of bile and gallbladder wall specimens.

INTERVENTIONS:
Other: Microbiological and histopathological investigation of bile and gallbladder wall specimens. — Bile and gallbladder wall specimens will be taken from all patients included in the study. The material will be sent for microbiological and histopathological investigation.

SUMMARY:
The aim of this project is to investigate the presence of bacteria in the gallbladder wall and the bile in patients undergoing cholecystectomy, to determine if the standard empirical antibiotic treatment used currently is effective against the most common pathogens.

DETAILED DESCRIPTION:
The investigators will compare two groups of patients; patients with acute calculous cholecystitis undergoing acute laparoscopic cholecystectomy and patients without cholecystitis undergoing elective laparoscopic cholecystectomy.

Secondly, the investigators wish to investigate if the presence of bacteria correlates with the grade of inflammation, and whether this can predict when cholecystitis is caused by infection.

In a clinical setting, this can provide important knowledge regarding the choice of antibiotics currently used to treat and prevent infection in the gallbladder.

The investigators will conduct two studies, one investigating the bacteria in bile and in the gallbladder wall and the resistens of the bacteria to antibiotics and another study investigating the histopathology of the gallbladder wall to see if the bacteria present is the cause of inflammation or an actual infection.

ELIGIBILITY:
Inclusion Criteria:

* Age above 18 years
* Signed consent form
* Patients having cholecystectomy performed at the Department of Surgery, Sygehus Lillebælt, Kolding.

Exclusion Criteria:

* Administration of any type of antibiotics one month prior to surgery in the control group.
* Previous instrumentation of the bileducts
* Previous clinical acute cholecystitis treated conservatively with antibiotics

Patients will be precluded from the studypopulation in cases of pPerioperative perforation of the gallbladder, or conversion to open cholecystectomy or in cases of failed attempts to extract bile or samples from the gallbladder wall.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The following data will be collected for all included patients:
  * Age
  * Sex
  * Weight
  * Height
  * BMI
  * Smoking
  * Alcohol
  * Diabetes
  * Cardiovascular disease
  * Preoperative blood samples
  * Use of antibiotic within the last year - what type and duration of treatment
  * Number of days with symptoms prior to the cholecystectomy
  * Vitals (blood pressure, pulse, saturation, respiratory rate, temperature)
  * Blood culture prior to the procedure in the case group
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Bacterial colonization in bile and gallbladder wall samples | 36-72 hours
  Microbiological investigation of microorganisms present in the bile and in the gallbladder wall.
  Bile samples will be collected by puncturing the gallbladder either perioperatively or immediate after extraction of the gallbladder from the abdomen. This is done in a sterile manner using a syringe.
  The gallbladder wall specimens are collected immediately after extraction of the gallbladder from the abdomen. Three samples will be taken from macroscopic normal looking parts of the posterior wall in the fundus area using a sterile 4 mm punch biopsy.
  Bile samples and punch biopsies sent to the Department of Clinical Microbiology, SLB, will be cultured on selected agar growth media and incubated under aerobic, microaerophilic, and anaerobic conditions.
  Bacterial colonies will be identified and quantified using routine laboratory methods.
Antibiotic resistans | 36-72 hours
  Microbiological investigation of antibiotic resistans of the bacteria, if any, present in bile and gallbladder wall specimens.
  Antimicrobial susceptibility testing will be performed using the disk diffusion method.
  To determine the possible presence of inhibitory concentrations of antibiotics in the bile samples, a droplet of bile from each sample will be added to an agar plate inoculated with the E. coli ATCC 25922-strain. After incubation, the appearance of a growth inhibition zone will be measured.
Histopathology of the gallbladder | 3-21 days
  Histopathological investigation of the gallbladder to investigate if there is either inflammation or an actual infection and correlate these findings to the bacterial colonization.
  The gallbladder from all included patients will be sent to the Department of Pathology, SLB, for evaluation of the grade of inflammation.
  After formalin fixation sections from the cystic duct, the corpus and the fundus area will be sampled. The sections will be embedded in paraffin and will be cut into thin slices, which will be dyed with hematoxylin and eosin. The grade of acute inflammation will be assessed in a semi quantitative manner:
  Grade 1: superficial ulceration of the mucosa concomitant with light infiltration by neutrophile granulocytes Grade 2: infiltration by granulocytes, spreading into the deeper layers of the gallbladder wall.
  Grade 3: profound necrosis, extending through the entire gallbladder wall.

CONTACTS AND LOCATIONS:
Overall Officials: Malene B Dissing, MD, Principal Investigator — Organkirurgisk afdeling, sygehus lillebælt, Kolding
Locations (1):
- Sygehus Lillebælt, Kolding, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kimura Y, Takada T, Kawarada Y, Nimura Y, Hirata K, Sekimoto M, Yoshida M, Mayumi T, Wada K, Miura F, Yasuda H, Yamashita Y, Nagino M, Hirota M, Tanaka A, Tsuyuguchi T, Strasberg SM, Gadacz TR. Definitions, pathophysiology, and epidemiology of acute cholangitis and cholecystitis: Tokyo Guidelines. J Hepatobiliary Pancreat Surg. 2007;14(1):15-26. doi: 10.1007/s00534-006-1152-y. Epub 2007 Jan 30. PMID 17252293
- [Background] Indar AA, Beckingham IJ. Acute cholecystitis. BMJ. 2002 Sep 21;325(7365):639-43. doi: 10.1136/bmj.325.7365.639. No abstract available. PMID 12242178
- [Background] Halpin V. Acute cholecystitis. BMJ Clin Evid. 2014 Aug 20;2014:0411. PMID 25144428
- [Background] Lou MA, Mandal AK, Alexander JL, Thadepalli H. Bacteriology of the human biliary tract and the duodenum. Arch Surg. 1977 Aug;112(8):965-7. doi: 10.1001/archsurg.1977.01370080063010. PMID 195558
- [Background] Fukunaga FH. Gallbladder bacteriology, histology, and gallstones. Study of unselected cholecystectomy specimens in Honolulu. Arch Surg. 1973 Feb;106(2):169-71. doi: 10.1001/archsurg.1973.01350140033011. No abstract available. PMID 4346851
- [Background] Sianesi M, Berri T. [Bacteriological studies on the bile in different conditions of surgical interest]. Chir Ital. 1976 Aug;28(4):341-55. Italian. PMID 1009648
- [Background] Brody LA, Brown KT, Getrajdman GI, Kannegieter LS, Brown AE, Fong Y, Blumgart LH. Clinical factors associated with positive bile cultures during primary percutaneous biliary drainage. J Vasc Interv Radiol. 1998 Jul-Aug;9(4):572-8. doi: 10.1016/s1051-0443(98)70324-0. PMID 9684825
- [Background] Siegman-Igra Y, Schwartz D, Konforti N, Perluk C, Rozin RR. Septicemia from biliary tract infection. Arch Surg. 1988 Mar;123(3):366-8. doi: 10.1001/archsurg.1988.01400270106016. PMID 3341915
- [Background] Park JW, Lee JK, Lee KT, Lee KH, Sung YK, Kang CI. How to interpret the bile culture results of patients with biliary tract infections. Clin Res Hepatol Gastroenterol. 2014 Jun;38(3):300-9. doi: 10.1016/j.clinre.2014.02.005. Epub 2014 Mar 24. PMID 24674840
- [Background] Rupp C, Bode K, Weiss KH, Rudolph G, Bergemann J, Kloeters-Plachky P, Chahoud F, Stremmel W, Gotthardt DN, Sauer P. Microbiological Assessment of Bile and Corresponding Antibiotic Treatment: A Strobe-Compliant Observational Study of 1401 Endoscopic Retrograde Cholangiographies. Medicine (Baltimore). 2016 Mar;95(10):e2390. doi: 10.1097/MD.0000000000002390. PMID 26962768
- [Background] Suh SW, Choi YS, Choi SH, Do JH, Oh HC, Kim HJ, Lee SE. Antibiotic selection based on microbiology and resistance profiles of bile from gallbladder of patients with acute cholecystitis. Sci Rep. 2021 Feb 3;11(1):2969. doi: 10.1038/s41598-021-82603-8. PMID 33536564
- [Background] Capoor MR, Nair D, Rajni, Khanna G, Krishna SV, Chintamani MS, Aggarwal P. Microflora of bile aspirates in patients with acute cholecystitis with or without cholelithiasis: a tropical experience. Braz J Infect Dis. 2008 Jun;12(3):222-5. doi: 10.1590/s1413-86702008000300012. PMID 18839486
- [Background] Gipson KS, Nickerson KP, Drenkard E, Llanos-Chea A, Dogiparthi SK, Lanter BB, Hibbler RM, Yonker LM, Hurley BP, Faherty CS. The Great ESKAPE: Exploring the Crossroads of Bile and Antibiotic Resistance in Bacterial Pathogens. Infect Immun. 2020 Sep 18;88(10):e00865-19. doi: 10.1128/IAI.00865-19. Print 2020 Sep 18. PMID 32661122
- [Background] Kwon W, Jang JY, Kim EC, Park JW, Han IW, Kang MJ, Kim SW. Changing trend in bile microbiology and antibiotic susceptibilities: over 12 years of experience. Infection. 2013 Feb;41(1):93-102. doi: 10.1007/s15010-012-0358-y. Epub 2012 Nov 21. PMID 23180506
- [Background] Begley M, Gahan CG, Hill C. The interaction between bacteria and bile. FEMS Microbiol Rev. 2005 Sep;29(4):625-51. doi: 10.1016/j.femsre.2004.09.003. PMID 16102595
- [Background] Ganzle MG, Hertel C, van der Vossen JM, Hammes WP. Effect of bacteriocin-producing lactobacilli on the survival of Escherichia coli and Listeria in a dynamic model of the stomach and the small intestine. Int J Food Microbiol. 1999 Apr 1;48(1):21-35. doi: 10.1016/s0168-1605(99)00025-2. PMID 10375132
- [Background] Maseda E, Maggi G, Gomez-Gil R, Ruiz G, Madero R, Garcia-Perea A, Aguilar L, Gilsanz F, Rodriguez-Bano J. Prevalence of and risk factors for biliary carriage of bacteria showing worrisome and unexpected resistance traits. J Clin Microbiol. 2013 Feb;51(2):518-21. doi: 10.1128/JCM.02469-12. Epub 2012 Nov 28. PMID 23196362
- [Background] Fisher K, Phillips C. The ecology, epidemiology and virulence of Enterococcus. Microbiology (Reading). 2009 Jun;155(Pt 6):1749-1757. doi: 10.1099/mic.0.026385-0. Epub 2009 Apr 21. PMID 19383684
- [Background] Arnold RS, Thom KA, Sharma S, Phillips M, Kristie Johnson J, Morgan DJ. Emergence of Klebsiella pneumoniae carbapenemase-producing bacteria. South Med J. 2011 Jan;104(1):40-5. doi: 10.1097/SMJ.0b013e3181fd7d5a. PMID 21119555
- [Background] van Dijk AH, de Reuver PR, Tasma TN, van Dieren S, Hugh TJ, Boermeester MA. Systematic review of antibiotic treatment for acute calculous cholecystitis. Br J Surg. 2016 Jun;103(7):797-811. doi: 10.1002/bjs.10146. Epub 2016 Mar 30. PMID 27027851
- [Background] Galili O, Eldar S Jr, Matter I, Madi H, Brodsky A, Galis I, Eldar S Sr. The effect of bactibilia on the course and outcome of laparoscopic cholecystectomy. Eur J Clin Microbiol Infect Dis. 2008 Sep;27(9):797-803. doi: 10.1007/s10096-008-0504-8. Epub 2008 Mar 28. PMID 18369670
- [Background] Grande M, Torquati A, Farinon AM. Wound infection after cholecystectomy. Correlation between bacteria in bile and wound infection after operation on the gallbladder for acute and chronic gallstone disease. Eur J Surg. 1992 Feb;158(2):109-12. PMID 1350211
- [Background] Adachi T, Eguchi S, Muto Y. Pathophysiology and pathology of acute cholecystitis: A secondary publication of the Japanese version from 1992. J Hepatobiliary Pancreat Sci. 2022 Feb;29(2):212-216. doi: 10.1002/jhbp.912. Epub 2021 Mar 27. PMID 33570821
- [Background] Panni RZ, Chatterjee D, Panni UY, Robbins KJ, Liu J, Strasberg SM. Sequential histologic evolution of gallbladder inflammation in acute cholecystitis over the first 10 days after onset of symptoms. J Hepatobiliary Pancreat Sci. 2023 Jun;30(6):724-736. doi: 10.1002/jhbp.1274. Epub 2022 Dec 1. PMID 36399043
- [Background] Mazeh H, Mizrahi I, Dior U, Simanovsky N, Shapiro M, Freund HR, Eid A. Role of antibiotic therapy in mild acute calculus cholecystitis: a prospective randomized controlled trial. World J Surg. 2012 Aug;36(8):1750-9. doi: 10.1007/s00268-012-1572-6. PMID 22456803
- [Background] Coccolini F, Sartelli M, Catena F, Montori G, Di Saverio S, Sugrue M, Ceresoli M, Manfredi R, Ansaloni L; CIAO and CIAOW Study Groups. Antibiotic resistance pattern and clinical outcomes in acute cholecystitis: 567 consecutive worldwide patients in a prospective cohort study. Int J Surg. 2015 Sep;21:32-7. doi: 10.1016/j.ijsu.2015.07.013. Epub 2015 Jul 17. PMID 26192973
- [Background] Jimenez E, Sanchez B, Farina A, Margolles A, Rodriguez JM. Characterization of the bile and gall bladder microbiota of healthy pigs. Microbiologyopen. 2014 Dec;3(6):937-49. doi: 10.1002/mbo3.218. Epub 2014 Oct 21. PMID 25336405
- [Background] Antimicrobial Resistance Collaborators. Global burden of bacterial antimicrobial resistance in 2019: a systematic analysis. Lancet. 2022 Feb 12;399(10325):629-655. doi: 10.1016/S0140-6736(21)02724-0. Epub 2022 Jan 19. PMID 35065702